CLINICAL TRIAL: NCT02027350
Title: Pressure-Volume Analysis of Constrictive Pericarditis
Brief Title: New Methods to Diagnose Constrictive Pericarditis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: due lack of subjects
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Barry Borlaug, Associate Professor of Medicine, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-008074
Record Dates: First submitted 2013-12-31; First posted 2014-01-06 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Constrictive Pericarditis
MeSH Terms: conditions — Pericarditis, Constrictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pressure-volume relationship (Experimental): Changes in pressure-volume relationships will be compared to changes in LV and RV systolic pressure during respiration.
  Interventions: Device: CD Leycom/Millar Instruments conductance catheter

INTERVENTIONS:
Device: CD Leycom/Millar Instruments conductance catheter — Conductance catheter-Pressure volume relationship

SUMMARY:
Until now, diagnosis of constriction was based on pressure changes of ventricle by conventional pressure-wide hemodynamic evaluation but not on ventricular volume change. This study will provide answers to persisting questions about volume changes during respiration in patients with constrictive pericarditis by directly measuring both right and left ventricular volume.

ELIGIBILITY:
Subjects referred for right and left heart catheterization will be eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Presence of constrictive pericarditis | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Barry Borlaug, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States